CLINICAL TRIAL: NCT05585905
Title: The Effect of Virtual Reality on the Behavior of Pediatric Dental Patients During Dental Sealant Application.
Brief Title: Virtual Reality in Pediatric Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Alexander Alcaaz, Principal Investigator, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UP-21-00583
Record Dates: First submitted 2022-10-12; First posted 2022-10-19 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Behavior, Child; Anxiety, Dental
Keywords: Virtual Reality; Dental; Local Anesthesia; Nitrous Oxide; Anxiety; Pain
MeSH Terms: conditions — Child Behavior; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Virtual Reality (Experimental): The virtual reality system being used for research purposes is the RelievRx by AppliedVR which is an immersive virtual reality device that includes a goggle headset and remote control. The VR experience will be an immersive experience where the child will interact with the system and navigate their way through a game that will involve bright colors, cartoon-like characters, and settings with age-appropriate content.
  Interventions: Device: Virtual Reality
- Basic Behavior Guidance Techniques (Active Comparator): The control sample will include basic behavior guidance techniques and is standard of care. The use of basic behavior guidance techniques is common in pediatric dentistry and is not unique to this study.
  Interventions: Behavioral: Basic Behavior Guidance Techniques

INTERVENTIONS:
Device: Virtual Reality — The VR system will be worn for approximately 5-10 minutes during dental sealant application
  Arms: Virtual Reality
Behavioral: Basic Behavior Guidance Techniques — Basic behavior guidance techniques will be used as a distraction technique when the VR system is not used during the dental sealant application
  Arms: Basic Behavior Guidance Techniques

SUMMARY:
Dental Fear and Anxiety is an emotional experiences affecting many children and adolescents which can lead to behavioral problems in the dental setting. The purpose of the proposed study is to investigate the effect of virtual reality on anxiety, behavior, and pain in children undergoing restorative dental procedures. Children enrolled in the study will include patients ages 6-18 who are healthy and require two or more dental sealants (at least one sealant per side). The participants in the study will serve as their own control using a split-mouth cross-over randomized control clinical trial design and will be randomly assigned to receive virtual reality or traditional behavior guidance techniques first during dental sealant placement. The objectives of this study are to explore the associations between the use of virtual reality distraction during dental sealant placement with Frankl score, FLACC scale, and anxiety based on the change in heart rate, and pain based on self-reported FPS-R when compared with to the control group. The crossover design will be assessed by a linear mixed model with patient treated as a random effect. This model will include treatment, visit, treatment by visit interaction term as well as a treatment sequence variable. Prior to analysis, the primary outcome measures will be assessed for normality using a Shapiro-Wilk statistic as well as quantile-quantile (QQ) plots. Should the data deviate sharply from a normal distribution, normalizing transformations will be sought and applied to the data.

DETAILED DESCRIPTION:
This study is a randomized controlled trial with a crossover design. Patients who are visiting the clinic for a comprehensive or periodic dental exam and are found to require two or more dental sealants (at least one sealant per side). The study subjects will include children ages 6-18 who are ASA I or II, as defined by the American Society of Anesthesiologists classification system. The proposed sample size for the study is 40 participants.

The children who are enrolled in the study will serve as both the experimental group and their own control. This is a split mouth design in which children who are enrolled in the study will serve as both the experimental group and their own control. After the child and parent are scheduled for the dental sealant appointment, they will be randomly assigned to receive the virtual reality system as a distraction technique for the first half or the latter half of the appointment (for research purposes). During the time when virtual reality is not used, traditional basic behavior guidance techniques will be used, as is the standard of care.

The virtual reality system being used for research purposes is the RelieVR by Applied VR which includes the goggle headset only. The VR experience will be an immersive experience where the child will interact with the system and navigate their way through a game that will involve bright colors, cartoon-like characters and settings with age-appropriate content. The VR system will be worn for approximately 5-10 minutes during the dental sealant application.

The dental sealant appointment will be video recorded, for research purposes and data collection. The video camera will be placed to include the child's face in order to monitor their facial expressions, legs movement, and activity during the administration of local anesthesia. The video camera will also be placed to include the blood pressure monitor and heart rate readings.

The behavior, pain, and anxiety will be analyzed at specific steps of the procedure including:

* Baseline (patient sitting in the chair prior to treatment)
* During sealant placement with Virtual Reality distraction
* During sealant placement with basic behavior guidance techniques
* Post Operative (patient sitting upright in chair, 5 minutes after procedure)

The Face, Legs, Activity, Cry, Consolability (FLACC) scale is a behavioral pain scale that will be conducted at the previously mentioned time intervals.

The patient's anxiety will be evaluated with a change in heart rate.

Additionally, at the end of each appointment for the duration of the study, the provider will assign the patient a Frankl behavior score 1-5, and record it in the patient's chart, as is the standard of care. The provider will also complete a Healthcare Provider Questionnaire through Qualtrics.

Data will be analyzed statistically to assess the relationship between a child's behavior (measured by the Frankl score and FLACCS scale), pain (measured by FPS-R), and anxiety (measured by heart rate) with the use of virtual reality or basic behavior guidance techniques.

The demographic factors will be collected from the patient's medical chart. The parent will be asked "how many hours of "screen time" (TV, computer, video games, tablet use), would you say that your child is allowed per week?". Parents and patients will also be asked to complete a satisfaction survey post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18
* ASA I or II
* Present to the Herman Ostrow School of Dentistry Pediatric Dental Clinic and Children's Dental Health Clinic at Long Beach Memorial Hospital for an initial or periodic exam, and are determined to require two or more dental sealants (at least one sealant per half mouth)

Exclusion Criteria:

Children with visual, auditory, or tactile deficits that would interfere with the ability to complete the experimental tasks

* Children who are unable to tolerate the RelievRx by AppliedVR will be screened after consenting to research participation by trying on the VR goggles and stating that they are comfortable and willing to proceed with wearing them during their dental appointment.
* Examples of children who may be unable to tolerate the VR goggles may include:

  * Children who wear glasses and are unable to comfortably adjust the system over their glasses
  * Children who experience dizziness, motion sickness or other discomfort during use
* Children who remove the VR goggles prior to dental sealant application
* Children who require pharmacological means to complete dental treatment (nitrous oxide, sedative drugs or general anesthesia)
* Children with a significant medical history of seizure disorders as flickering from devices can trigger epileptic episodes.
* Children with developmental disabilities
* Children with a psychiatric disorder, organic brain syndrome, mental retardation, or other known cognitive/neurological disorders
* Children that are not English or Spanish speaking

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-17 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in behavior on the FLACCS scale | Baseline, Immediately after sealant placement with Virtual Reality, Immediately after sealant placement with basic behavior guidance techniques
  Behavior Rating Score (FLACCS): Patient's behavior as rated by the FLACC behavioral pain scale.
  FLACC score includes facial expressions, leg movement, activity (bodily movement), crying, and consolability. Each category is score on the 0-2 scale resulting in a in a total score of 0-10.
  * 0 = Relaxed and comfortable
  * 1-3 = Mild discomfort
  * 4-6 = Moderate pain 12
  * 7-10 = Severe discomfort/pain
Change in behavior on the FRANKL Scale | Baseline, IImmediately after sealant placement with Virtual Reality, Immediately after sealant placement with basic behavior guidance techniques, and immediately after completion of dental treatment
  Patient's behavior as rated by the dental provider within one of the following categories: 1= definitely negative, 2= negative, 3= positive, 4= definitely positive. This scale is routinely used by dentists and documented in the patient chart.
Change in anxiety | Baseline, Immediately after sealant placement with Virtual Reality, Immediately after sealant placement with basic behavior guidance techniques, and immediately after completion of dental treatment
  Measured by change in heart rate (eg. beats per minute)
Patient perceived pain | Immediately after sealant placement with Virtual Reality, Immediately after sealant placement with basic behavior guidance techniques
  Patient's pain will be evaluated using the self-assessment Face Pain Scale- Revised (FPS-R) taken at outlined points (above) during restorative procedure.
  The FPS-R has 0-to-10 metric. The scale shows a close linear relationship with visual analog pain scales. Score the chosen face 0, 2, 4, 6, 8, or 10, counting left to right, so "0" equals "No pain" and "10" equals "Very much pain."

SECONDARY OUTCOMES:
Parent Satisfaction | 5 minutes after the completion of treatment
  Will be evaluated post treatment for the Virtual Reality and standard of care. Satisfaction questions will be asked on a scale on a scale of 1 to 10.
Patient Satisfaction | 5 minutes after the completion of treatment
  Will be evaluated post treatment for the Virtual Reality and standard of care. Satisfaction questions will be asked on a scale on a scale of 1 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Angela Alvarez, DMD, Study Chair — Herman Ostrow School of Dentistry Pediatric Department
Locations (2):
- United States (2):
  - Children's Dental Health Clinic, Long Beach, California
  - Herman Ostrow School of Dentistry Pediatric Department, Los Angeles, California

REFERENCES:
- [Background] Sharma A, Kumar D, Anand A, Mittal V, Singh A, Aggarwal N. Factors predicting Behavior Management Problems during Initial Dental Examination in Children Aged 2 to 8 Years. Int J Clin Pediatr Dent. 2017 Jan-Mar;10(1):5-9. doi: 10.5005/jp-journals-10005-1397. Epub 2017 Feb 27. PMID 28377646
- [Background] Cianetti S, Lombardo G, Lupatelli E, Pagano S, Abraha I, Montedori A, Caruso S, Gatto R, De Giorgio S, Salvato R. Dental fear/anxiety among children and adolescents. A systematic review. Eur J Paediatr Dent. 2017 Jun;18(2):121-130. doi: 10.23804/ejpd.2017.18.02.07. PMID 28598183
- [Background] Ramos-Jorge ML, Marques LS, Pavia SM, Serra-Negra JM, Pordeus IA. Predictive factors for child behaviour in the dental environment. Eur Arch Paediatr Dent. 2006 Dec;7(4):253-7. doi: 10.1007/BF03262561. PMID 17164071
- [Background] Porritt J, Marshman Z, Rodd HD. Understanding children's dental anxiety and psychological approaches to its reduction. Int J Paediatr Dent. 2012 Nov;22(6):397-405. doi: 10.1111/j.1365-263X.2011.01208.x. Epub 2012 Jan 3. PMID 22221141
- [Background] Moore R, Brodsgaard I. Dentists' perceived stress and its relation to perceptions about anxious patients. Community Dent Oral Epidemiol. 2001 Feb;29(1):73-80. PMID 11153566
- [Background] American Academy of Pediatric Dentistry. Behavior guidance for the pediatric dental patient. The Reference Manual of Pediatric Dentistry. Chicago, Ill.: American Academy of Pediatric Dentistry; 2021:306-24.
- [Background] Aminabadi NA, Farahani RM, Balayi Gajan E. The efficacy of distraction and counterstimulation in the reduction of pain reaction to intraoral injection by pediatric patients. J Contemp Dent Pract. 2008 Sep 1;9(6):33-40. PMID 18784857
- [Background] Khandelwal M, Shetty RM, Rath S. Effectiveness of Distraction Techniques in Managing Pediatric Dental Patients. Int J Clin Pediatr Dent. 2019 Jan-Feb;12(1):18-24. doi: 10.5005/jp-journals-10005-1582. PMID 31496566
- [Background] Lopez-Valverde N, Muriel Fernandez J, Lopez-Valverde A, Valero Juan LF, Ramirez JM, Flores Fraile J, Herrero Payo J, Blanco Antona LA, Macedo de Sousa B, Bravo M. Use of Virtual Reality for the Management of Anxiety and Pain in Dental Treatments: Systematic Review and Meta-Analysis. J Clin Med. 2020 Apr 5;9(4):1025. doi: 10.3390/jcm9041025. PMID 32260538 (Retraction: PMID 32731319 J Clin Med. 2020 Jul 28;9(8):)
- [Background] Piskorz J, Czub M. Effectiveness of a virtual reality intervention to minimize pediatric stress and pain intensity during venipuncture. J Spec Pediatr Nurs. 2018 Jan;23(1). doi: 10.1111/jspn.12201. Epub 2017 Nov 20. PMID 29155488
- [Background] Walther-Larsen S, Petersen T, Friis SM, Aagaard G, Drivenes B, Opstrup P. Immersive Virtual Reality for Pediatric Procedural Pain: A Randomized Clinical Trial. Hosp Pediatr. 2019 Jul;9(7):501-507. doi: 10.1542/hpeds.2018-0249. Epub 2019 Jun 3. PMID 31160472
- [Background] Li A, Montano Z, Chen VJ, Gold JI. Virtual reality and pain management: current trends and future directions. Pain Manag. 2011 Mar;1(2):147-157. doi: 10.2217/pmt.10.15. PMID 21779307
- [Background] Carl E, Stein AT, Levihn-Coon A, Pogue JR, Rothbaum B, Emmelkamp P, Asmundson GJG, Carlbring P, Powers MB. Virtual reality exposure therapy for anxiety and related disorders: A meta-analysis of randomized controlled trials. J Anxiety Disord. 2019 Jan;61:27-36. doi: 10.1016/j.janxdis.2018.08.003. Epub 2018 Aug 10. PMID 30287083
- [Background] Lahti S, Suominen A, Freeman R, Lahteenoja T, Humphris G. Virtual Reality Relaxation to Decrease Dental Anxiety: Immediate Effect Randomized Clinical Trial. JDR Clin Trans Res. 2020 Oct;5(4):312-318. doi: 10.1177/2380084420901679. Epub 2020 Jan 21. PMID 31962052
- [Background] Tanja-Dijkstra K, Pahl S, White MP, Andrade J, May J, Stone RJ, Bruce M, Mills I, Auvray M, Gabe R, Moles DR. Can virtual nature improve patient experiences and memories of dental treatment? A study protocol for a randomized controlled trial. Trials. 2014 Mar 22;15:90. doi: 10.1186/1745-6215-15-90. PMID 24655569
- [Background] Hosey MT, Blinkhorn AS. An evaluation of four methods of assessing the behaviour of anxious child dental patients. Int J Paediatr Dent. 1995 Jun;5(2):87-95. doi: 10.1111/j.1365-263x.1995.tb00170.x. PMID 7547819
- [Background] American Academy of Pediatric Dentistry. Use of nitrous oxide for pediatric dental patients. The Reference Manual of Pediatric Dentistry. Chicago, Ill.: American Academy of Pediatric Dentistry; 2020:324-9.
- [Background] Merkel SI, Voepel-Lewis T, Shayevitz JR, Malviya S. The FLACC: a behavioral scale for scoring postoperative pain in young children. Pediatr Nurs. 1997 May-Jun;23(3):293-7. PMID 9220806
- [Background] Hockenberry MJ, Wilson D, Winkelstein ML: Wong's Essentials of Pediatric Nursing, ed, 7, St Louis, 2005 p.1259. Used with permission. © Mosby